CLINICAL TRIAL: NCT00922116
Title: A Single Arm, Open Label Study to Assess the Efficacy, Safety and Tolerability of Once-monthly Administration of Subcutaneous Mircera® for the Maintenance of Haemoglobin Levels in Patients With Chronic Renal Anaemia Who Are Not on Dialysis
Brief Title: A Study of Once Monthly Subcutaneous Mircera in Patients With Chronic Renal Anemia Not on Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22285
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — sc every month (starting dose of 100, 120, 150 or 200 micrograms based on previous ESA therapy)

SUMMARY:
This single arm study will assess the efficacy, safety and tolerability of once monthly administration of subcutaneous Mircera for the maintenance of hemoglobin levels in patients with chronic renal anemia not on dialysis.Patients will receive sc Mircera at a starting dose of 100, 120, 200 or 360 micrograms every 4 weeks, calculated from the last weekly dose of ESA previously administered. Subsequent doses will be adjusted to maintain hemoglobin levels within the target range. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* chronic renal anemia;
* continuous maintenance ESA therapy with the same dosing interval during the previous month, and no change in totally weekly dose.

Exclusion Criteria:

* transfusion of red blood cells during previous 2 months;
* poorly controlled hypertension;
* significant acute or chronic bleeding;
* active malignant disease (except non-melanoma skin cancer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2009-04-30 (Actual); Primary Completion 2010-11-30 (Actual); Study Completion 2010-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- South Korea (10):
  - Inje University Busan Paik Hospital; Nephrology, Busan
  - Kyungpook National Uni Hospital; Internal Medicine, Daegu
  - Chungnam National Uni Hospital; Nephrology, Daejeon
  - Chonnam National University Hospital, Gwangju
  - NHIC Ilsan Hospital, Kyonggi-do
  - Seoul National Uni Hospital; Internal Medicine, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Severance Hospital; Division of Nephrology, Seoul
  - East-West Neo Medical Center; Division Of Nephology, Seoul
  - Samsung Medical Centre; Department of Hematology & Oncology, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera: Participants received Mircera (methoxy polyethylene glycol epoetin beta) at a starting dose of 120, 200 or 360 micrograms [mcg] (based on previous erythropoiesis stimulating agent therapy) administered via subcutaneous (SC) injection once monthly for 24 weeks. Doses were titrated based on hemoglobin levels.
Period: Overall Study
Arm/Group | Mircera
Started | 191
Completed | 176
Not Completed | 15
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: Safety population defined as all participants who participated in the trial.
Groups:
- Mircera: Participants received Mircera (methoxy polyethylene glycol epoetin beta) at a starting dose of 120, 200 or 360 mcg (based on previous erythropoiesis stimulating agent therapy) administered via SC injection once monthly for 24 weeks. Doses were titrated based on hemoglobin levels.
Arm/Group | Mircera
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114
  Male | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Average Hemoglobin Concentration Within the Target Range During the Efficacy Evaluable Period (EEP)
Description: The target hemoglobin was defined as the mean of the three assessments recorded at Weeks -4, -2, and 0 (Stability Verification Period [SVP]). EEP was an 8 week period from Weeks 17 to 24. The 95 percent (%) confidence interval (CI) was estimated using Clopper-Pearson.
Time Frame: EEP (Weeks 17 to 24)
Population: Intention-to-Treat (ITT) population included all participants who received one more dose of Mircera.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 187
percentage of participants | 53.9 [46.3 to 61.4]

2. Secondary Outcome: Change in Hemoglobin Concentration Between SVP and the EEP
Description: Baseline hemoglobin was defined as the mean of the three assessments recorded at Weeks -4, -2, and 0 (SVP). EEP hemoglobin was defined as the mean of the hemoglobin assessments during EEP. EEP was an 8 week period from Weeks 17 to 24.
Time Frame: SVP (Baseline), and EEP (Weeks 17 to 24)
Population: ITT population.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Mircera
Number analyzed (Participants) | 187
grams per deciliter (g/dL) | 0.55 (0.93)

3. Secondary Outcome: Percentage of Participants Maintaining Hemoglobin Concentration Within Hemoglobin Range 10.0 to 12.0 g/dL Throughout the EEP
Description: EEP was an 8 week period from Weeks 17 to 24. The 95% CI was estimated using Clopper-Pearson.
Time Frame: EEP (Weeks 17 to 24)
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 187
percentage of participants | 73.0 [65.9 to 79.4]

4. Secondary Outcome: Percentage of Participants Who Required Dose Adjustments During Dose Titration Period (DTP) and EEP
Description: DTP was a 16- week period from Week 1 to Week 16, EEP was an 8-week period from Weeks 17 to 24. Dose adjustment was assessed during entire Week 1 to 24.
Time Frame: Weeks 1 to 24
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera
Number analyzed (Participants) | 187
percentage of participants | 87.2

5. Secondary Outcome: Time Spent in Hemoglobin Range of 10.0 to 12.0 g/dL During DTP and EEP
Description: as for outcome 4
Time Frame: Weeks 1 to 24
Population: ITT population. Here number of participants analyzed = participants who were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mircera
Number analyzed (Participants) | 158
days | 103.6 (41.9)

6. Secondary Outcome: Average Dose of Mircera Per Month
Time Frame: Weeks 0-4, 4-8, 8-12, 12-16, 16-20, and 20-24
Population: ITT population. Here number of participants analyzed = participants who were analyzed for the outcome measure.
Measure: Mean (Standard Deviation); unit: microgram (mcg)
Arm/Group | Mircera
Number analyzed (Participants) | 145
microgram (mcg)
  Week 0-4 | 121.2 (9.8)
  Week 4-8 | 100.8 (33.3)
  Week 8-12 | 78.8 (45.8)
  Week 12-16 | 72.7 (46.6)
  Week 16-20 | 66.9 (48.0)
  Week 20-24 | 66.2 (47.1)

ADVERSE EVENTS:
Time Frame: up to Week 28
Arm/Group | Mircera
Serious Adverse Events (participants affected / at risk) | 31/191
Other Adverse Events (participants affected / at risk) | 90/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=191)
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Glaucoma (Eye disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Generalised oedema (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Gout (Metabolism and nutrition disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Diabetic nephropathy (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera (N=191)
Oedema (General disorders) | 16
Nasopharyngitis (Infections and infestations) | 17
Upper respiratory tract infection (Infections and infestations) | 20
Hyperkalaemia (Metabolism and nutrition disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 10
Hypertension (Vascular disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.